CLINICAL TRIAL: NCT05496699
Title: The Comparsion of MCkenzie and Mulligan Exercise in Patients With Non-Specific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstinyeFTR
Record Dates: First submitted 2022-02-07; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Neck Pain
Keywords: neck pain; exercise; manuel therapy; physiotherapy
MeSH Terms: conditions — Neck Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: 2 group, intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mckenzie group (Experimental): Mckenzie exercise protocol will be applied to the participants in this group. It will be applied to the participants for 4 weeks and 5 days a week for 30 minutes. The exercise program will be performed by the patient under the supervision of a physiotherapist.
  Interventions: Behavioral: Mckenzie Exercises
- mullgian group (Experimental): Mulligan exercise protocol will be applied to the participants in this group. It will be applied to the participants for 4 weeks and 5 days a week for 30 minutes. The exercise program will be performed by the patient under the supervision of a physiotherapist.
  Interventions: Behavioral: Mulligan Exercise

INTERVENTIONS:
Behavioral: Mckenzie Exercises — 1. Cervical Retraction Exercise in Sitting Position The participant sits on the chair, puts the second and third fingers on his chin and pushes his head posteriorly and inferiorly.
  2. Cervical Rotation Exercise in Sitting Position
  3. Cervical Retraction Exercise in Supine Position
  4. Cervical Rotation Exercise in Supine Position The participant turns his head to the right and left, respectively, while taking his head back in the supine position with his head out of the bed.
  5. Cervical Lateral Flexion Exercise
  6. Cervical Flexion Exercise in Sitting Position
  Arms: mckenzie group
Behavioral: Mulligan Exercise — The exercises to be applied are listed below.
  1- C1-C2 Self Mobilization Slip is applied for natural apophyseal cervical right rotation. The belt is put on level C1. At the same time, the participant actively pulls the belt and turns his head to the right. To facilitate the rotation of the belt in C1, pressure is applied to the belt in the same direction as C2 and rotation of the head towards the restricted side is requested. It waits like this for 3 seconds. These movements are done in the painless range.
  Arms: mullgian group

SUMMARY:
Non-specific neck pain (NSBA) is defined as pain in the posterior and lateral parts of the neck in the absence of neurological and specific pathologies (fracture, infection, inflammation, etc.) between the superior nuchael line and the 1st thoracic vertebra. The lifetime neck pain rate is approximately 12-70%; Neck pain is the reason for admission in approximately 25% of applications to outpatient clinics of the Physical Medicine and Rehabilitation Clinic. Neck pain is the most common spinal problem after low back pain, and it is defined as nonspecific neck pain due to its multifactorial etiology. Many conservative treatment methods are used in the treatment of NSBA. These include medical treatments, exercise, massage, acupuncture, neural therapy and physical therapy modalities. The basis of Mulligan's theory is based on a positional error that develops secondarily, causing misplacement of the joint. With the Mulligan mobilization technique, the joint is displaced to normal and positional error is corrected. Restoration of motion is aimed by repositioning the bone. The main indication in this technique is increased pain, stiffness and weakness in movement. The Mulligan mobilization technique is performed by asking for active movement while maintaining a manually applied joint shift. Painless movement is aimed at the joint. According to the general principles of Mulligan treatment, all techniques are applied in a way that does not cause pain and creates an effect that will eliminate the pain in a short time after the application.

DETAILED DESCRIPTION:
The McKenzie approach is an evaluative and therapeutic strategy in the practice of musculoskeletal physiotherapy to manage pain and restore the function of the cervical spine. This approach aims to control cervical disability when used in the early stages such as postural correction and increasing flexibility of adjacent musculotendinous structures. It aims to classify mechanically induced spinal pain into postural, dysfunctional and dysregulation syndromes to centralize and reduce spinal pain. Cervical self-treatment techniques used by McKenzie specialists have been shown to be effective for nonspecific neck pain. The purpose of evaluating patients with cervical-related disorders is to select self-management techniques as directional preference movements that should be repeated to reduce pain and symptoms. When we look at the studies in the literature; It has been reported that Mulligan concept techniques improve pain and disability symptoms in patients with chronic mechanical neck pain at the short- and medium-term effect level. In a study comparing Mulligan and McKenzie practices previously, it was concluded that Mulligan exercise was more effective in improving cervical range of motion than McKenzie exercise in adults with reduced cervical lordosis. In another comparative article, according to the results of the study comparing the two exercise techniques, it was seen that cervical ROM increased in both exercise groups.

However, it was concluded that the Mulligan exercise group showed better results than the Mckenzie group in the early period. Different types of mobilization are used to treat neck pain, but limited studies have been conducted to compare the effectiveness of two different mobilization techniques in the treatment of neck pain.

The aim of the study was that two different exercise programs (mckenzi-mulligan) were used in individuals with non-specific neck pain; to compare their effects on pain, range of motion (ROM) and functional outcomes. It is aimed to compare the effect of Mulligan exercises and Mckenzie exercises on pain reduction, joint range of motion, recovery speed, muscle activation and functional treatment in individuals with non-specific neck pain due to non-specific neck pain due to multifactorial etiology. Considering that there should be a larger number of studies on this subject with the literature review, it is aimed to contribute this study to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with neck pain of unknown origin for more than 3 months
* Individuals between the ages of 18-45
* Non-smokers
* Individuals who have the ability to understand and apply Turkish written and verbal instructions

Exclusion Criteria:

* Individuals with a history of neck injury, micro or macro trauma,
* Individuals with tumors in and around the spinal cord,
* Individuals who have undergone surgery from the neck and shoulder region,
* Individuals with positive Vertebrobacillary Artery Test,
* Female individuals who are pregnant, individuals receiving hormone therapy,
* Individuals with neurological disease,
* Individuals with neuropathic pain due to neurological and systemic disorders,
* Patients with any loss of function in the upper extremities due to musculoskeletal disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | First week
  A visual analog scale will be used to assess participants' degree of neck pain before and after treatment. It will be created by marking the instantaneous pain according to the levels on a scale with the visual analog scale. The pain felt by the person will be marked as "0: no pain", "10: I feel very severe pain". Scoring will be made from the parts marked on the plane over the points given by the person. The validity and reliability study of the scale was done by Price et al. made by The scale was adapted to Turkish by A. Aydın et al.
Neck Disability Index | First week
  In order to evaluate neck functionality, Vernon et al. Developed by Turkish version study Aslan et al. made by The Neck Disability Questionnaire includes a total of 10 questions such as pain, personal care, concentration, working, driving, and sleeping. Each question will be scored between 0-5 points. The survey will be evaluated out of a maximum of 50 points. 0 points means no restrictions, 50 points means full apology. 0-4 points will be considered as no disability, 5-14 points as mild disability, 14-24 points as moderate disability, 25-34 points as severe disability and 35 and above as complete disability.

SECONDARY OUTCOMES:
Evaluation of Muscle Strength | First week
  A hand held dynamometer, which is a valid and reliable method, will be used to evaluate muscle strength. (17) Neck muscle strength will be evaluated in four directions with extension, forward flexion, and right and left lateral flexion. The position of the dynamometer will be adjusted at the occipital protuberance for extension, above the eyebrows for forward flexion, and above the corresponding ear for right lateral flexion and left lateral flexion. The tests will be repeated three times and patients will be given a rest period of at least one minute between repetitions. The highest value from the results obtained with these measurements will be recorded in Newton (N) as the maximum force to be used in statistical analysis.
Tampa Kinesiophobia Scale | First week
  17-question survey will be conducted to assess participants' injury avoidance and fear of movement. The scale is scored with Likert scoring (1 = I strongly disagree, 4 = I completely agree). The total score is between 17-68, and it is understood that the higher the score the participant gets, the higher the kinesiophobia. A total score of more than 37 is considered as a high degree of kinesiophobia. (20)
Fremantle Neck Awareness Questionnaire | First week
  Fremantle Neck Awareness Questionnaire will be applied to the participants in order to evaluate the relationship between kinesiophobia and neck awareness. Likert type assessing individual-specific altered perception (0 = Never/Never feel this way, 1 = I rarely feel this way, 2 = Sometimes, or sometimes I feel this way, 3 = I feel this way often, 4 = I feel this way all or most of the time) It's a simple survey. The questionnaire asks individuals 9 questions such as how they perceive their neck relative to their body, how they perceive their body position.
Corbin Posture Analysis | First week
  Corbin Posture Analysis For posture assessment, Corbin et al.'s form was used, in which postural disorders were scored according to severity (0=absent, 1=mild, 2=moderate, 3=well-severe) by observing the case from the lateral and posterior.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Pamukçu, Principal Investigator — Istinye University
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No